CLINICAL TRIAL: NCT02990286
Title: Evaluation of Efficacy and Safety of Rituximab in Association With Mycophenolate Mofetil Versus Mycophenolate Mofetil Alone in Patients With Interstitial Lung Diseases (ILD) Non-responders to a First-line Immunosuppressive Treatment
Brief Title: Evaluation of Efficacy and Safety of Rituximab With Mycophenolate Mofetil in Patients With Interstitial Lung Diseases
Acronym: EvER-ILD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRN15-SMA/EvER-ILD
Record Dates: First submitted 2016-11-25; First posted 2016-12-13 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lung Disease, Interstitial
Keywords: Non specific intertitial pneumonia; interstitial pneumonia with autoimmune feature; connective tissue disease; rituximab; Mycophenolate Mofetil; pulmonary fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases; Pulmonary Fibrosis | interventions — Rituximab; Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab with Mycophenolate Mofetil (Experimental)
  Interventions: Drug: Rituximab; Drug: Mycophenolate Mofetil
- Placebo of rituximab with Mycophenolate Mofetil (Placebo Comparator)
  Interventions: Drug: Placebo of Rituximab; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Rituximab — Rituximab 500mg concentrate for solution for infusion. One course of IV rituximab consisting of a first infusion of 1000 mg (500 ml solution) rituximab (day 1 infusion), and a second infusion of 1000 mg (500 ml solution) rituximab two weeks later (day 15 infusion)
  Arms: Rituximab with Mycophenolate Mofetil
Drug: Placebo of Rituximab — 500 ml of saline (0.9% sodium chloride) for infusion One course of intravenous placebo of rituximab consisting of a first infusion of 500 ml of saline (0.9% sodium chloride) infusion (day 1 infusion), and a second infusion of 500 ml of saline infusion two weeks later (day 15 infusion)
  Arms: Placebo of rituximab with Mycophenolate Mofetil
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 500mg film-coated tablets
  1 gram twice daily on oral route of MMF (= 2 grams daily) for 6 months.

SUMMARY:
The purpose of the study is to evaluate the efficacy on lung function 6 months after one course of rituximab (2 infusions) and mycophénolate mofétil (MMF) treatment compared to one course of placebo and 6 months of MMF treatment in a broad range of patients with Interstitial Lung Diseases (ILD) non-responders to a first line immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. A diagnosis of ILD:

   * ILD associated with differentiated CTD or IPAF (based on internationally accepted criteria)
   * OR idiopathic ILD
3. A diagnosis of NSIP based on:

   * a histological pattern of NSIP
   * OR HRCT findings suggestive of NSIP defined as basal predominant reticular abnormalities with traction bronchiectasis, peri-bronchovascular extension and subpleural sparing, frequently associated with ground-glass attenuation
4. Patients who did not respond or relapsed or were not able to continue at least one first-line immunosuppressive treatment of ILD: corticosteroids, azathioprine, cyclophosphamide or other immunosuppressants. For the assessment of clinical response, the absence of response was defined as: either a decrease or an increase, but <10% in % predicted FVC.
5. Subjects covered by or having the rights to French social security (including CMU),
6. Written informed consent obtained from subject, with a specific check box on the Consent form of the study, understanding the risk for men and women treated with mycophenolate mofetil. And additional written consent from subject on the care and contraception agreement form for women of childbearing potential treated with mycophenolate.
7. Ability for subject to comply with the requirements of the study

Exclusion Criteria:

1. Known diagnosis of significant respiratory disorders (asthma, tuberculosis, sarcoidosis, aspergillosis, or cystic fibrosis) other than CTD-NSIP, IPAF-NSIP and iNSIP
2. Evidence of any clinically significant, severe or unstable, acute or chronically progressive cardiac (severe heart failure New York Heart Association Class IV or severe uncontrolled cardiac disease), other medical disease (other than NSIP) or surgical disorder, or any condition that may affect patient safety in the judgment of the investigator.
3. HRCT pattern of typical usual interstitial pneumonia (UIP)
4. For patients with idiopathic ILD, HRCT pattern of possible UIP (no evocative of NSIP)
5. Histological pattern other than pattern of NSIP
6. A first line treatment with MMF or rituximab
7. Known hypersensitivity to MMF or rituximab or sulfonamide antibiotics
8. Treatment with immunosuppressive treatments other than corticosteroids:

   * azathioprine, cyclophosphamide, methotrexate, cyclosporine, tacrolimus, leflunomide within 2 weeks (5 half-lives <= 2 weeks) prior to inclusion
   * intravenous immunoglobulins, hydroxychloroquine or other monoclonal antibody therapies (such as but not limited to etanercept, adalimumab, efalizumab, infliximab, golimumab, certolizumab) within 6 months (5 half-lives <= 6 months) prior to inclusion
9. Patients registered on a pulmonary transplantation list
10. Patients with known hypoxanthine-guanine phosphoribosyl-transferase (HGPRT) hereditary deficiency (such as Lesch-Nyhan and Kelley-Seegmiller syndrome)
11. Pregnant or breastfeeding women, or women of child-bearing potential not using two reliable contraceptive methods (including female partners of sexually active men treated with mycophenolate) and men not using a contraceptive method (condom), or women and men having a pregnancy project during the year following randomization.
12. Patients at significant risk for infectious complications: HIV positive, other known immunodeficiency syndromes, untreated tuberculosis, hepatitis B and C or other known viral infection, infection requiring anti-infectious treatment in the preceding 4 weeks
13. Current history of substance and/or alcohol abuse
14. Deprivation of liberty, under judicial protection
15. Participation in another biomedical research with experimental drug or medical device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Change in FVC in % of predicted | From baseline to 6 months
  Change in FVC (in % of predicted) since declines in FVC correlates with increased risk of subsequent mortality in ILD patients and FVC is one of the core set of outcomes defined in interstitial lung diseases. Data obtained from the two groups of patients (rituximab and placebo) will be compared to each other. FVC will be performed in each study center in a standardized manner according to the ATS/ERS recommendations and ECCS reference equations

SECONDARY OUTCOMES:
Progression Free Survival (PFS). | PFS measured at 3, 6 and 12 months
  PFS is defined as the time 1) to the first acute exacerbation, or 2) to an absolute decline of 10 % points in the percentage of the predicted FVC, or 3) to the necessity to withdraw the MMF with/without a new immunosuppressive treatment (except corticoids), or 4) to death or 5) registration to a lung transplantation list. An acute exacerbation is defined by (1) progressive dyspnea over 1 month or less; (2) new pulmonary infiltrates on chest radiography or computed tomography, and (3) the absence of an overt underlying cause of rapid deterioration
Changes in the quality of life score | Changes from baseline to 6 months in the quality of life score, and, changes from baseline to 6 months in the visual analogic scales of dyspnea and cough
  The quality of life score as measured by the SF-36 v1.3 questionnaire, version developed and validated in interstitial lung disease (ILD) patients.
Changes in the visual analogic scales of dyspnea | Changes from baseline to 6 months in the quality of life score, and, changes from baseline to 6 months in the visual analogic scales of dyspnea and cough
  Changes in the visual analogic scales of dyspnea (EVA test)
Cough evaluation | Changes from baseline to 6 months in cough evaluation
  Changes in cough evaluation
Cumulative doses of corticoids for the 2 groups | Cumulative doses of corticoids at 6 months
  Cumulative doses of corticoids for the 2 groups
Changes in the FVC expressed as % of predicted | Changes from baseline to 3 and 6 months in the FVC expressed as % of predicted
  Changes in the FVC expressed as % of predicted
Changes in DLCO | Changes from baseline to 6 months in DLCO
  Changes in DLCO
Changes in the 6-minutes-walk test | Changes from baseline to 6 months in the 6-minutes-walk test
  Changes in the 6-minutes-walk test
Changes in autoantibodies concentration | Changes from baseline to 6 months in autoantibodies concentration
  Changes in autoantibodies concentration
Changes in biological markers related to lymphocyte B depletion: CD19 lymphocytes | Changes from baseline to 6 months in lymphocytes B CD19
  Changes in biological markers related to lymphocyte B depletion: CD19 lymphocytes
Changes in gammaglobulins | Changes from baseline to 6 months in gammaglobulins
  Changes in gammaglobulins
Changes in HRCT of the chest images | Changes from baseline to 6 months in HRCT of the chest images
  Changes in HRCT of the chest images
Adverse events related to treatment | Adverse events during the 6 months of study period
  In particular infectious adverse events and biological blood disorders during the 6 months of study period will be collected
Rituximab PK parameters : distribution volume | Points at Day1, Day15, 3 and 6 months
  Rituximab PK parameters : distribution volume
Rituximab clearance | Points at Day1, Day15, 3 and 6 months
  Rituximab clearance
Half-life of rituximab in blood | Points at Day1, Day15, 3 and 6 months
  Half-life of rituximab in blood

CONTACTS AND LOCATIONS:
Overall Officials: TRACLET Julie, Principal Investigator — HC LYON; NUNES Hilario, Principal Investigator — AP-HP - Hôpital Avicenne; CRESTANI Bruno, Principal Investigator — AP-HP - Hôpital Bichat; ISRAEL BIET Dominique, Principal Investigator — AP-HP HEGP; NACCACHE Jean-Marc, Principal Investigator — AP-HP - Hôpital Tenon; WEMEAU Lidwine, Principal Investigator — CHRU LILLE; JOUNEAU Stéphane, Principal Investigator — CHU Rennes; PREVOT Grégoire, Principal Investigator — University Hospital, Toulouse; REYNAUD-GAUBERT Martine, Principal Investigator — AP-HM Hôpital Nord; HIRSCHI SANTELMO Sandrine, Principal Investigator — CHRU Strasbourg; GONDOUIN Anne, Principal Investigator — Centre Hospitalier Universitaire de Besancon; COURT-FORTUNE Isabelle, Principal Investigator — CHU ST-ETIENNE; BONNIAUD Philippe, Principal Investigator — CHU DIJON; QUETANT Sébastien, Principal Investigator — University Hospital, Grenoble; GOMEZ Emmanuel, Principal Investigator — CHU NANCY; BLANC François-Xavier, Principal Investigator — Nantes University Hospital; MARQUETTE Charles-Hugo, Principal Investigator — CHU NICE; MARCHAND-ADAM Sylvain, Principal Investigator — CHRU TOURS
Locations (5):
- France (5):
  - Chu Besancon, Besançon
  - Chu Dijon, Dijon
  - AP-HM Hôpital NORD, Marseille
  - Chu Rennes, Rennes
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mankikian J, Caille A, Reynaud-Gaubert M, Agier MS, Bermudez J, Bonniaud P, Borie R, Brillet PY, Cadranel J, Court-Fortune I, Crestani B, Debray MP, Gomez E, Gondouin A, Hirschi-Santelmo S, Israel-Biet D, Jouneau S, Juvin K, Leger J, Kerjouan M, Marquette CH, Naccache JM, Nunes H, Plantier L, Prevot G, Quetant S, Traclet J, Valentin V, Uzunhan Y, Wemeau-Stervinou L, Bejan-Angoulvant T, Cottin V, Marchand-Adam S; EVER-ILD investigators and the OrphaLung network. Rituximab and mycophenolate mofetil combination in patients with interstitial lung disease (EVER-ILD): a double-blind, randomised, placebo-controlled trial. Eur Respir J. 2023 Jun 8;61(6):2202071. doi: 10.1183/13993003.02071-2022. Print 2023 Jun. PMID 37230499
- [Derived] Bejan-Angoulvant T, Naccache JM, Caille A, Borie R, Nunes H, Ferreira M, Cadranel J, Crestani B, Cottin V, Marchand-Adam S; OrphaLung. Evaluation of efficacy and safety of rituximab in combination with mycophenolate mofetil in patients with nonspecific interstitial pneumonia non-responding to a first-line immunosuppressive treatment (EVER-ILD): A double-blind placebo-controlled randomized trial. Respir Med Res. 2020 Nov;78:100770. doi: 10.1016/j.resmer.2020.100770. Epub 2020 May 23. PMID 32777737